CLINICAL TRIAL: NCT06938672
Title: Evaluating the Effects of tDCS on Sleep and Cognition in Healthy Older Adults: A Randomised Controlled Trial Using a Nap Design
Brief Title: Evaluating the Effects of tDCS on Sleep and Cognition in Healthy Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-6636-10284
Record Dates: First submitted 2025-03-13; First posted 2025-04-22 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Sleep; Cognition; Healthy Aging
Keywords: sleep; healthy aging; cognition; tDCS; non-invasive brain stimulation; nap
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transcranial Direct Current Stimulation (tDCS) (Active Comparator): Transcranial direct current stimulation. Participants will experience a 20-minute session of active tDCS (1.2 mA) on two consecutive days.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Placebo Transcranial Direct Current Stimulation (tDCS) (Placebo Comparator): Transcranial direct current stimulation. Participants will experience a 20-minute session of placebo tDCS on two consecutive days.
  Interventions: Device: Placebo Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Placebo Transcranial Direct Current Stimulation (tDCS) — Placebo Transcranial direct current stimulation (tDCS): Participants will experience a 20-minute session of placebo tDCS on two consecutive days.
  Other Names: sham tDCS
  Arms: Placebo Transcranial Direct Current Stimulation (tDCS)
Device: Active Transcranial Direct Current Stimulation (tDCS) — Active transcranial direct current stimulation (tDCS). Participants will experience a 20-minute session of active tDCS (1.2 mA) on two consecutive days.
  Other Names: tDCS
  Arms: Active Transcranial Direct Current Stimulation (tDCS)

SUMMARY:
The goal of this interventional study is to learn if transcranial direct current stimulation (tDCS), a gentle, cost-effective and non-invasive brain stimulation technique can improve sleep brain activity during an afternoon nap. Since these sleep brain patterns are linked to better memory, attention, and thinking skills, this study aims to find out if improving sleep in a nap can also enhance these cognitive skills in healthy older adults (aged 60+).

The main questions it aims to answer are:

* Can a short (20-minute) tDCS session before a nap improve sleep patterns during the nap?
* Since these sleep patterns are linked to memory and attention, can tDCS also improve thinking skills after the nap?
* Are two tDCS session more effective than one for improving nap sleep and thinking skills?

Participants will:

• Be required to come to the university for testing over four days.

During each session they will:

* Complete computer based-tasks to assess memory and thinking.
* Receive a 20-minute session of either real (active) or fake (placebo) tDCS.
* Take a short, monitored nap while researchers measure sleep activity (using polysomnography - a gold-standard, non-invasive sleep monitoring tool).
* Complete an easy-to-use sleep test at home on the nights after the naps.

  * Wear a lightweight watch (called an Actiwatch) throughout the study period to track sleep and movement.
  * Complete daily sleep diaries.

By taking part, participants will help researchers understand whether tDCS can improve sleep during naps and, in turn, support memory and thinking skills. This research could lead to better treatments for sleep problems, help protect brain health, and reduce the risk of dementia as people age. The brain stimulation in this study may also help improve their sleep and cognition.

DETAILED DESCRIPTION:
Sleep is vital for maintaining physical and cognitive health across the lifespan. However, normal age-related changes to sleep can impair memory, learning, and waste clearance in the brain, contributing to the risk of cognitive decline and dementia.

Transcranial direct current stimulation (tDCS), a non-invasive technique that modulates brain activity, shows promise for enhancing both sleep and cognition. However, existing studies have significant methodological limitations. Notably, very few have investigated 'offline' tDCS -where stimulation is applied before sleep- to assess objective sleep changes using polysomnography (PSG). Instead, most research has relied on subjective measures, consistently finding that offline tDCS enhances perceived sleep quality, especially with repeated stimulation sessions. Importantly, offline tDCS may be more feasible for use outside laboratory settings compared to 'online' approaches, where stimulation is applied during sleep, making it a more scalable intervention.

Furthermore, delivering tDCS before a daytime nap, rather than nocturnal sleep, offers additional advantages by reducing participant burden, particularly in older adults. Studies applying tDCS during a nap in older adults have shown improvements in objective sleep microstructure and declarative memory. By contrast, studies applying tDCS during nocturnal sleep have reported inconsistent results. Despite its potential benefits, no studies have explored the effects of an offline, nap-based tDCS approach on objective sleep outcomes.

Additionally, few studies have examined whether repeated sessions of offline tDCS might amplify its effects on objective PSG-measured sleep. While repeated sessions have been shown to positively influence subjective sleep outcomes, it remains unclear whether the same benefits apply to objective sleep metrics. This study will address this gap by investigating whether two sessions of offline tDCS, compared to one, are necessary to improve objective sleep outcomes.

In summary, this study aims to determine whether offline tDCS applied prior to a nap can enhance objective sleep during a daytime nap and improve post-nap cognitive performance in older adults. If effective, this low-burden, non-invasive intervention could serve as a practical tool for promoting healthy aging and reducing dementia risk.

The primary objectives of this randomised, placebo-controlled crossover trial are:

To evaluate the impact of offline tDCS on objective sleep microstructure and architecture during naps.

To assess the effects of tDCS on post-nap cognitive performance. To examine the cumulative effect of two tDCS sessions upon objective sleep and cognition, compared to one.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60+ years
* Speak fluent English
* Be cognitively healthy
* A self-reported good sleeper, with a regular sleep pattern

Exclusion Criteria:

* The presence of any major physical or psychiatric illness or comorbidities
* Self-reported neurodegenerative dementia or other neurological disorders
* Self-reported relevant sleep disorders or disturbances
* Those with irregular sleep schedules (i.e. night shift workers)
* A PSQI score above 5 (as this is associated with significant sleep disturbance)
* Relevant skin allergies
* Taking medication that affects the central nervous system or sleep, or consume caffeine, alcohol or cigarettes excessively
* Metallic or electronic implants

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Sleep spindle density | During nap immediately after tDCS application
  PSG-measured slow (11.99 - 12.99Hz) and fast (13 - 14.99Hz) sleep spindle density
Sleep spindle amplitude | During nap immediately after tDCS application
  PSG-measured slow (11.99 - 12.99Hz) and fast (13 - 14.99Hz) sleep spindle amplitude
Slow wave sleep amplitude | During nap immediately after tDCS application
  PSG-measured SWS amplitude (peak-to-peak, μV)
Slow wave sleep density | During nap immediately after tDCS application
  PSG-measured slow wave sleep density (number of slow waves divided by the minutes of sleep)
Verbal declarative memory | Baseline (before tDCS/nap) and 15 minutes after the nap
  Change in Verbal Paired Associates Word Learning Task performance will be measured by % correct recall at baseline (before the tDCS intervention and nap) compared to % correct recall 15 minutes after the nap has taken place.
Attentional Network Task (ANT) | Baseline (before tDCS/nap) and 15 minutes after the nap
  Change in Attentional Network Task performance will be measured by Reaction Time (RT) (Milliseconds (ms) at baseline (before the tDCS intervention and nap) compared to RT (ms) 15 minutes after the nap has taken place.
Attentional Network Task (ANT) | Baseline (before tDCS/nap) and 15 minutes after the nap
  Change in Attentional Network Task performance will be measured by Accuracy (%) at baseline (before the tDCS intervention and nap) compared to Accuracy (%) 15 minutes after the nap has taken place.

SECONDARY OUTCOMES:
Visuo-spatial declarative picture memory | Baseline (before tDCS/nap) and 15 minutes after the nap
  Change in Picture Memory performance will be measured by Accuracy (% Correct) at baseline (before the tDCS intervention and nap) compared to Accuracy (% Correct) 15 minutes after the nap has taken place.
Visuo-spatial declarative location memory | Baseline (before tDCS/nap) and 15 minutes after the nap
  Change in Location Memory performance will be measured by Accuracy (% Correct) at baseline (before the tDCS intervention and nap) compared to Accuracy (% Correct) 15 minutes after the nap has taken place

CONTACTS AND LOCATIONS:
Overall Officials: Rosie H Musgrave, BA Hons, RPSGT, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No